CLINICAL TRIAL: NCT05961059
Title: Phase Ia/b Double-blind, Placebo-controlled, Dose Escalating Safety Study of Detoxified Shigella Flexneri 2a Artificial Invasin Complex (InvaplexAR-Detox) Vaccine Formulated with and Without DmLT Adjuvant Given Intramuscularly to Healthy Adults in the Netherlands and Zambia
Brief Title: InvaplexAR-Detox and DmLT Adjuvant in the Netherlands and Zambia
Acronym: SUNSHINE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Centre for Infectious Disease Research in Zambia (Other); PATH (Other); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); Göteborg University (Other); European Vaccine Initiative (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Principal Investigator, Meta Roestenberg, Priniciple Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: SUNSHINE
Record Dates: First submitted 2023-07-05; First posted 2023-07-27 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Shigellosis; Bacillary Dysentery
Keywords: Vaccine; Invaplex; dmLT; Shigella
MeSH Terms: conditions — Dysentery, Bacillary

STUDY DESIGN:
Intervention Model Description: A phase Ia/b dose escalation, randomized, double-blind, placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- A1 - Low dose vaccine (Netherlands) (Experimental): 10 Dutch participants who receive three 2.5 μg doses of the vaccine without adjuvant at a 28-day interval in Cohort A.
  Interventions: Biological: 2.5 μg InvaplexAR-Detox
- A2 - Low dose vaccine + adjuvant (Netherlands) (Experimental): 10 Dutch participants who receive three 2.5 μg dose of the vaccine with 0.1 μg of adjuvant at a 28-day interval in Cohort A.
  Interventions: Biological: 2.5 μg InvaplexAR-Detox; Biological: 0.1 μg of dmLT
- B1/C1 - High dose vaccine (Netherlands & Zambia) (Experimental): 10 Dutch participants who receive three 10 μg vaccine doses without adjuvant at a 28-day interval in Cohort B and 15 Zambian participants who receive three 10 μg vaccine doses without adjuvant at a 28-day interval in Cohort C.
  Interventions: Biological: 10 μg InvaplexAR-Detox
- B2/C2 - High dose vaccine + adjuvant (Netherlands & Zambia) (Experimental): 10 Dutch participants that receive three 10 μg vaccine doses with 0.1 μg of adjuvant at a 28-day interval in Cohort B and 15 Zambian participants that receive three 10 μg vaccine doses with 0.1 μg of adjuvant at a 28-day interval in Cohort C.
  Interventions: Biological: 10 μg InvaplexAR-Detox; Biological: 0.1 μg of dmLT
- A3/B3/C3 - Placebo (Netherlands & Zambia) (Placebo Comparator): 5 Dutch participants who receive three placebo vaccinations at a 28-day interval in Cohort A, another 5 Dutch participants who receive three placebo vaccinations at a 28-day interval in Cohort B and 5 Zambian participants who receive three placebo vaccinations at a 28-day interval in Cohort C.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: 2.5 μg InvaplexAR-Detox — 2.5 μg intramuscular dose of Sfl2a InvaplexAR-Detox.
  Arms: A1 - Low dose vaccine (Netherlands); A2 - Low dose vaccine + adjuvant (Netherlands)
Biological: 10 μg InvaplexAR-Detox — 10 μg intramuscular dose of Sfl2a InvaplexAR-Detox.
  Arms: B1/C1 - High dose vaccine (Netherlands & Zambia); B2/C2 - High dose vaccine + adjuvant (Netherlands & Zambia)
Biological: 0.1 μg of dmLT — 0.1 μg intramuscular dose of double mutant (LT R192G/L211A) enterotoxigenic Escherichia coli heat labile toxin (dmLT).
  Arms: A2 - Low dose vaccine + adjuvant (Netherlands); B2/C2 - High dose vaccine + adjuvant (Netherlands & Zambia)
Biological: Placebo — Placebo vaccination with commercially available saline solution.
  Arms: A3/B3/C3 - Placebo (Netherlands & Zambia)

SUMMARY:
The goal of this clinical trial is to test a new Shigella vaccine (InvaplexAR-DETOX) in combination with a new adjuvant (dmLT) in healthy participants. The main questions it aims to answer are:

* Is the new Shigella vaccine (with and without the new adjuvant) safe and well tolerated?
* How wel does the new Shigella vaccine stimulate the immune system in combination with the new adjuvant, and without the new adjuvant?

Participants will receive three vaccinations at 28-day intervals. Researchers will compare the results of participants vaccinated with the vaccine in combination with the adjuvant to the results of participants vaccinated with the vaccine only and to the results of participants vaccinated with a placebo (fake vaccine).

DETAILED DESCRIPTION:
Rationale: Shigella remains endemic in many places and occurs in epidemics that cause considerable morbidity and mortality. Vaccines are an attractive and potentially highly cost-effective tool for the prevention of shigellosis and can fill current gaps in effective prevention strategies. A challenge to effective Shigella vaccine development has been the reduced immunogenicity and protective efficacy of candidate Shigella vaccines in infants and children less than 3 years of age. The potential impact of including an adjuvant in candidate parenteral Shigella vaccine formulations needs to be evaluated. InvaplexAR-Detox is an injectable Shigella vaccine that uses a novel combination of conserved invasion plasmid antigen proteins with a serotype-specific bacterial lipopolysaccharide attenuated for safe intramuscular administration. The adjuvant dmLT has been shown to significantly enhance Shigella immune responses in mice and has safely been administered intramuscularly in healthy volunteers in combination with other antigens in phase I trials.

Objective: to evaluate the safety and immunogenicity of two strength formulations of a candidate Shigella vaccine (2.5 or 10 μg Sfl2a InvaplexAR-Detox) given with and without adjuvant (0.1 μg dmLT).

Study design: this is a phase Ia/b dose escalation, randomized, double-blind, placebo-controlled trial assessing the safety, tolerability and immunogenicity of three vaccinations given 4 weeks apart of Sfl2a InvaplexAR-Detox vaccine alone or in combination with the dmLT adjuvant in the Leiden University Medical Center in the Netherlands and at the Centre for Infectious Disease Research in Zambia (CIDRZ). The study will be initiated with the low vaccine dose in the Netherlands (Cohort A) and will not proceed to the high vaccine dose in the Netherlands (Cohort B) before the safety data of Cohort A has been reviewed by the Safety Monitoring Committe (SMC). The SMC will also review the safety data of Cohort B before the high vaccine dose will be administered in Zambian adults (Cohort C).

Study population: a total of 50 healthy Dutch and 35 healthy Zambian adults aged 18-50 years.

Intervention: a 2.5 μg or 10 μg intramuscular dose of the candidate Shigella vaccine Sfl2a InvaplexAR-Detox given with and without double mutant (LT R192G/L211A) enterotoxigenic Escherichia coli heat labile toxin adjuvant (0.1 μg dmLT) given at day 1, day 29 and day 57 compared to a placebo (saline).

Main study endpoints: Primary endpoint measures are the occurrence of solicited and unsolicited adverse events considered to be related to vaccination. Secondary outcome measures are humoral and cellular immune responses to vaccination with and without adjuvant compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult, male or female, aged 18 to 50 years (inclusive) at the time of inclusion (=vaccination).
2. Provide written informed consent before initiation of any study procedures.
3. Available to complete all study visits and procedures.
4. Negative stool PCR test for Shigella.
5. Women of childbearing potential: negative pregnancy test at screening and before each study vaccine administration. Women are considered not of childbearing potential if they are postmenopausal (no menses for 12 months without an alternative medical cause), or if they have no uterus or no ovaries. Women of childbearing potential must agree to use continuous adequate contraception to avoid pregnancy during the study, for at least 4 weeks before the first vaccination and for 3 months following the last vaccine dose.

Adequate methods of contraception for this study include:

1. hormonal contraception

1. combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal)
2. progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or implantable) 2. intrauterine device (IUD) 3. intrauterine hormone-releasing system (IUS) 4. bilateral tubal occlusion/litigation procedure 5. vasectomized partner (the vasectomized partner should be the sole male sexual partner for that participant).

   6. sexual abstinence (defined as refraining from heterosexual intercourse from signing the informed consent until 3 months after the last vaccine dose).
   1. Any history or evidence of clinically relevant chronic medical conditions (such as: psychiatric conditions, diabetes mellitus, hypertension [treated by medication], autoimmune disorders, immunodeficiencies, cardiovascular, renal disease or inflammatory bowel disease). Trial physicians (in consultation with the principal investigator) will use clinical judgement on a case-by-case basis to assess safety risks under this criterion.
   2. Current use of immunosuppressive medications (except for antihistamines and topical or inhalation corticosteroids).
   3. Women who are a) currently nursing or b) who are pregnant or planning to become pregnant during the study period plus 3 months beyond the last vaccine dose.
   4. Participation in research involving another investigational product (defined as receipt of an investigational product or exposure to an invasive investigational device) 30 days before the first vaccination or anytime through the last in-clinic study safety visit.
   5. Positive blood test for hepatitis B surface antigen (HbsAg), hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
   6. Clinically significant abnormalities on basic laboratory screening tests.
   7. Systemic antimicrobial treatment (i.e., topical treatments are not an exclusion criterion) within 1 week before the first vaccine dose (temporary exclusion).
   8. Known hypersensitivity to compounds in the vaccine or adjuvant or other known drug allergies that may increase the risk of adverse events.
   9. Regular use (weekly or more often) of antidiarrheal, anti-constipation, or antacid therapy.
   10. Abnormal stool pattern (fewer than 3 stools per week or more than 3 stools per day) on a regular basis; loose or liquid stools on other than an occasional basis.
   11. Personal or family history of inflammatory arthritis.
   12. Proven allergy to any substance in the InvaplexAR-Detox vaccine or dmLT or history of anaphylactic reaction to any other vaccine.
   13. Exclusionary skin disease history/findings that would confound assessment or prevent appropriate monitoring of local AEs, or possibly increase the risk of local AEs.
   14. Recent (<3 months) history of gastroenteritis.
   15. Received previous licensed or experimental Shigella vaccine, dmLT or live Shigella challenge.
   16. Any severe medical condition that might place the participant at increased risk of adverse events according to the clinical judgment of the study clinicians in consultation with the PI.
   17. Any planned vaccination within 14 days before the first vaccine dose until the last in-clinic study visit, with the exception of SARS-CoV-2 vaccines or influenza vaccines.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-identified male or female
Enrollment: 85 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Occurence of solicited adverse events | Within 7 days following vaccination (day of vaccination and 7 subsequent days).
  Occurrence of solicited adverse events considered to be (possibly, probably or definitely) related to vaccination according to the International Classification of Diseases version 11 (ICD-11) compared to the placebo group. Local solicited adverse events include pain/tenderness, erythema, induration/swelling, pruritus, and ipsilateral axillary lymphadenopathy. Systemic solicited adverse events include fever, chills, headache, fatigue, malaise, nausea/vomiting, painful/swollen joints, myalgia, diarrhea, and abdominal pain. Only symptoms with an onset after a vaccination until the 7th subsequent day after that vaccination will be considered solicited.
Occurence of unsolicited adverse events | Within 28 days following each vaccination (day of vaccination and 28 subsequent days).
  Occurrence of unsolicited adverse events considered to be (possibly, probably or definitely) related to vaccination, according to the ICD-11 classification.

SECONDARY OUTCOMES:
Geometric mean titers of serum immunoglobulin A antibodies to Invaplex antigens | Study days 1 (baseline), 29, 57, 64, 85 and 225.
  Serum GMTs of anti-LPS, anti-IpaB and anti-IpaC IgA
Geometric mean titers of serum immunoglobulin G antibodies to Invaplex antigens | Study days 1 (baseline), 29, 57, 64, 85 and 225.
  Serum GMTs of anti-LPS, anti-IpaB and anti-IpaC IgG
Proportion of participants with immunoglobulin A seroconversion (> 4-fold rise in titer over baseline) | Study days 1 (baseline), 29, 57, 64, 85 and 225.
  Percentage of participants wit a ≥ 4-fold increase in serum anti-LPS, anti-IpaB and anti-IpaC IgA titer from baseline
Proportion of participants with immunoglobulin G seroconversion (> 4-fold rise in titer over baseline) | Study days 1 (baseline), 29, 57, 64, 85 and 225.
  Percentage of participants wit a ≥ 4-fold increase in serum anti-LPS, anti-IpaB and anti-IpaC IgG titer from baseline
Serum bactericidal assay response to S. flexneri 2a, strain 2457T in geometric mean titers | Study days 1 (baseline), 29, 57, 64, and 85.
Proportion of participants with serum bactericidal assay responses (≥ 4-fold rise over baseline) to S. flexneri 2a, strain 2457T | Study days 1 (baseline), 29, 57, 64, and 85.
Geometric mean titers of α4β7 antibodies in lymphocyte supernatant. | Study days 1 (baseline), 8, 36, and 64
B cell memory responses to Invaplex antigens | Study days 1 (baseline), 64 and 225
  B cell memory responses to the LPS and IpaB and IpaC antigens.
T cell memory responses to Invaplex antigens | Study days 1 (baseline), 64 and 225
  T cell memory responses to the LPS and IpaB and IpaC antigens.

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data of the trial will follow the FAIR (findable, accessible, interoperable and re-usable) principles for data collection and sharing outlined by force11 and metadata will be entered in a repository which will be open access after completion of the trial.
Time Frame: After completion of the trial. Specific timepoint to be decided.

REFERENCES:
- [Derived] Roozen GVT, Sukwa N, Chirwa M, White JA, Estrada M, Maier N, Turbyfill KR, Laird RM, Suvarnapunya AE, Sayeh A, D'Alessio F, Marion C, Pattacini L, Hoogerwerf MA, Murugan R, Terrinoni M, Holmgren JR, Sirima SB, Houard S, Simuyandi M, Roestenberg M. Safety, Tolerability, and Immunogenicity of the InvaplexAR-DetoxShigella Vaccine Co-Administered with the dmLT Adjuvant in Dutch and Zambian Adults: Study Protocol for a Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Phase Ia/b Clinical Trial. Vaccines (Basel). 2025 Jan 8;13(1):48. doi: 10.3390/vaccines13010048. PMID 39852827